CLINICAL TRIAL: NCT03862625
Title: The Effect of a New-designed Modular Adaptive Seating System on Coronal and Sagittal Balance of the Spine and Pelvic Obliquity in Children With Nonambulatory Cerebral Palsy and Scoliosis
Brief Title: Seating System for Scoliosis in Non-ambulatory Children With Cerebral Palsy: A Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Damla Korkmaz (Other)
Responsible Party: Sponsor-Investigator, Merve Damla Korkmaz, Assistant doctor, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/72
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy; Neuromuscular Scoliosis
Keywords: cerebral palsy; scoliosis; adaptive seating system; sagittal balance; pelvic obliquity; coronal balance
MeSH Terms: conditions — Cerebral Palsy; Scoliosis

STUDY DESIGN:
Intervention Model Description: There are two groups in this study. In the first group, there is home exercises program for scoliosis and a modular adaptive seating system. In the second group there is only home exercises program for scoliosis. The nonambulatory children between the ages of 6-15 with cerebral palsy and scoliosis were randomly grouped according to the order of Pediatric Rehabilitation Unit of Istanbul University, Istanbul Faculty of Medicine, Physical Medicine and Rehabilitation Department.
Who Masked: Outcomes Assessor
Masking Description: In our clinical study, the person who performed radiographic evaluations before and after treatment did not know about the treatments received by the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a modular adaptive seating system (Experimental): In the first group, there is home exercises program for scoliosis and a modular adaptive seating system.
  Interventions: Device: a modular adaptive seating system; Other: home exercise program for scoliosis
- home exercises for scoliosis (Active Comparator): In the second group there is only home exercise program for scoliosis.
  Interventions: Other: home exercise program for scoliosis

INTERVENTIONS:
Device: a modular adaptive seating system
  Other Names: home exercise program for scoliosis
  Arms: a modular adaptive seating system
Other: home exercise program for scoliosis

SUMMARY:
The effect of a modular seating system on coronal and sagittal balance of the spine and pelvic obliquity in children with non-ambulatory (Gross Motor Function Classification System Level IV-V) and scoliosis

The hypothesis in our study is; a modular adaptive seating system prevents the progression of spinal curvature and Reimer's maturation index, improves the sagittal balance of the spine and pelvic obliquity.

DETAILED DESCRIPTION:
Aim: The aim of this study was to evaluate the effect of a modular adaptive seating system and exercise therapy for scoliosis on the progression of spinal curvature, spinal sagittal balance and pelvic obliquity in children aged 6 to 15 years with cerebral palsy (Gross Motor Function Classification System (GMFCS) level IV-V) and scoliosis.

Materials and methods: A prospective, randomized and controlled, single-blind study was performed on 29 patients with cerebral palsy(CP). Patients were randomized into two groups. Both groups were given scoliosis home exercise program at least three days a week and 10 repetitions for each exercise in a day. In the first group, a modular adaptive seating system used for at least four hours in a day with exercise program for scoliosis. This seating system includes a sitting elevation that corrects the pelvic obliquity, the hip block that prevents the sliding from the sitting floor and a body support unit that provides the alignment of the spine and controls of the body. Cobb angle, pelvic obliquity, sagittal spino-pelvic parameters (thoracic kyphosis angle (TK), lumbar lordosis angle (LL), sagittal vertical axis (SVA), pelvic tilt (PT), pelvic incidence (PI), sacral slop (SS)) and Reimer's migration index (RMI) measurements were evaluated by Surgimap® software at the before and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* the participant 6 to 15 years of age during inclusion
* the participant is diagnosed as cerebral palsy by a specialist
* the participant's Cobb angle is between 10-40 degrees. (Cobb angle above 40 degrees and patients whose parents have not accepted the operation)
* There is no history of operation due to scoliosis or the decision of the operation has not been accepted by the patients and their parents
* the participant is Gross Motor Function Classification System Level 4 or 5
* Lack of contracture to prevent sitting in the lower extremity
* Parents agree to participate in the intensive therapy program and stop the therapeutic interventions for scoliosis and lower extremities during the 3-month follow-up period

Exclusion Criteria:

* Having a history of operation due to scoliosis
* The deformity in the spine is rigid
* If the curvature measured in the spine is less than 10 degrees or more than 40 degrees in the patients whose operation decision is accepted by the family
* Having a seating modification applied at least 1 year before being included in the study
* Having a spasticity and contracture to prevent sitting in the hip and knee joint
* Having a pressure ulcer to prevent the patient from sitting
* the participant has comorbidity that is not related about cerebral palsy
* Having epileptic seizures not controlled
* Having bone operations for hip joints

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2019-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merve D Korkmaz, 1, Principal Investigator — Istanbul University; Murat Korkmaz, 2, Principal Investigator — Koc University Hospital; Resa Aydın, 3, Study Director — Istanbul University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It will be available for sharing after publication.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 nonambulatory children aged 6-15 years with CP and scoliosis who were admitted to Istanbul University, Istanbul Medical Faculty, Pediatric Rehabilitation Unit of the Department of Physical Medicine and Rehabilitation were included in the study
Groups:
- a Modular Adaptive Seating System: In the first group, there is home exercises program for scoliosis and a modular adaptive seating system.
  a modular adaptive seating system
  home exercise program for scoliosis
- Home Exercises for Scoliosis: In the second group there is only home exercise program for scoliosis.
  home exercise program for scoliosis
Period: Overall Study
Arm/Group | a Modular Adaptive Seating System | Home Exercises for Scoliosis
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | a Modular Adaptive Seating System | Home Exercises for Scoliosis | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 8 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 15 | 15 | 30
Gross Motor Function Classification System (GMFCS) [Count of Participants; unit: Participants] — The Gross Motor Function Classification System (GMFCS) is a 5 level classification system that describes the gross motor function of cerebral palsy on the basis of self-initiated movement abilities.
  GMCFS level I: Can walk indoors and outdoors and climb stairs without using hands for support.
  GMFCS level II:Can climb stairs with a railing GMFCS level III: Walks with assistive mobility devices indoors and outdoors on level surfaces GMFCS level IV: Walking ability severely limited even with assistive devices GMFCS level V: Has physical impairments that restrict voluntary control of movement
  Participants
    GMFCS level IV | 4 | 2 | 6
    GMFCS level V | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cobb Angle
Description: cobb angle shows the curvature of the spine in the coronal plane
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | a Modular Adaptive Seating System | Home Exercises for Scoliosis
Number analyzed (Participants) | 15 | 14
degrees | 23.77 (12.98) | 26.31 (9.99)

2. Primary Outcome: Pelvic Obliquity
Description: pelvic obliquity is posture of pelvis in relation to the ground
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | a Modular Adaptive Seating System | Home Exercises for Scoliosis
Number analyzed (Participants) | 15 | 14
degrees | 6.46 (3.15) | 7.39 (4.28)

3. Primary Outcome: Sagittal Balance
Description: sagittal balance of the spine is the posture of the spine on the sagittal plane
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | a Modular Adaptive Seating System | Home Exercises for Scoliosis
Number analyzed (Participants) | 15 | 14
degrees
  thoracal kyphosis | 33.75 (11.95) | 41.07 (9.97)
  lombar lordosis | 36.25 (9.90) | 36.16 (9.43)
  pelvic tilt | 20.99 (13.62) | 13.37 (7.86)
  sacral slope | 31.04 (14.93) | 31.84 (11.4)
  pelvic incidence | 52.4 (11.9) | 45.22 (11.34)
  Sagittal vertical axis (SVA) | 10.93 (7.46) | 13.48 (6.58)

4. Secondary Outcome: Reimer's Migration Index (RMI)
Description: it shows the degree of hip subluxation or dislocation
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of hip subluxation
Arm/Group | a Modular Adaptive Seating System | Home Exercises for Scoliosis
Number analyzed (Participants) | 15 | 14
percentage of hip subluxation
  RMI for right hip | 26.27 (11.20) | 22.85 (7.65)
  RMI for left hip | 39.80 (22.28) | 32.43 (9.70)

ADVERSE EVENTS:
Time Frame: 12 week-period
Description: The participants has been controlled for advers events. These are pressure ulsers on sitting surfaces and pain at the spinal muscles.
Arm/Group | a Modular Adaptive Seating System | Home Exercises for Scoliosis
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

LIMITATIONS AND CAVEATS:
First, the participants only in CP with GMCFS level V. Second, the short follow-up period can be counted could be selected as a limitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03862625/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2019-02-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03862625/SAP_000.pdf